CLINICAL TRIAL: NCT02745912
Title: A Phase 1, Open-Label, Sequential Design Study to Evaluate the Potential Effect of Multiple Oral Doses of Extended-Release Combination of Naltrexone and Bupropion on the Pharmacokinetics of a Single Oral Dose of Metformin in Healthy Subjects
Brief Title: Study to Evaluate the Effect of Naltrexone and Bupropion Combination on the Pharmacokinetics of Metformin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orexigen Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NaltrexBuprop-1004; U1111-1166-8630 (Registry Identifier: WHO)
Record Dates: First submitted 2016-04-18; First posted 2016-04-20 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Healthy Subjects
Keywords: Drug Therapy
MeSH Terms: interventions — Naltrexone; Bupropion; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin + Naltrexone/Bupropion (Experimental): Metformin (850 mg, immediate release tablet, orally, once on Day 1 and Day 14) naltrexone/bupropion (8/90 mg/mg, extended-release tablets, orally, twice daily from Day 3 through Day 5 and 16/180 mg/mg, twice daily from Day 6 through Day 15.
  Interventions: Drug: Naltrexone/Bupropion; Drug: Metformin

INTERVENTIONS:
Drug: Naltrexone/Bupropion — Naltrexone/Bupropion extended-release tablets.
Drug: Metformin — Metformin immediate-release tablet.

SUMMARY:
The purpose of this study is to determine the effect of multiple oral doses of naltrexone/bupropion on the pharmacokinetics (PK) of a single oral dose of metformin.

DETAILED DESCRIPTION:
The drug being tested in this study is naltrexone HCl and bupropion HCl Extended- Release fixed dose combination (NB) . This study will evaluate the potential effect of multiple oral doses of extended-release combination of naltrexone/bupropion on the PK of a single oral dose of metformin in healthy participants with normal renal function (defined as creatinine clearance [CrCl] greater than equal to [>=] 90 milliliter per minute [mL/min]/1.73 meter square [m^2]).

The study will enroll approximately 30 participants. Participants will receive:

Metformin 850 mg as a single dose alone and in combination with multiple doses of Naltrexone/Bupropion Naltrexone 8 mg/Bupropion 90 mg + Naltrexone 16 mg/Bupropion 180 mg as multiple doses alone and in combination with a single dose of metformin

All participants will be asked to take 1 tablet of metformin in the morning on Day 1 and Day 14, 1 tablet of naltrexone/bupropion twice daily from Day 3 through Day 5, and 2 tablets of naltrexone/bupropion twice daily from Day 6 through Day 15.

This single center trial will be conducted in the United States. The overall time to participate in this study is 73 days. Participants will be admitted on Day -1 (check in) and remain confined to the clinic until Day 16 and will be contacted by telephone 30 (±2) days after last dose of study drug for a follow-up assessment. Serial blood samples will be collected for PK assessments. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy male or female.
2. Is aged 18 to 55 years, inclusive, at signing of informed consent and first dose of study drug.
3. Weighs at least 50 kilogram (kg) and has a body mass index (BMI) of 18.0 to 40.0 kilogram per square meter (kg/m^2), inclusive, at Screening.
4. Has normal renal function (defined as CrCl >=90 mL/min/1.73 m^2) at Screening and Check-in (Day -1).
5. A female subject of childbearing potential* who is sexually active with a nonsterilized* male partner agrees to use adequate contraception* from signing of informed consent throughout the duration of the study and for 12 weeks after the last dose of study drug.

Exclusion Criteria:

1. Has known hypersensitivity to metformin, bupropion, naltrexone, or any component of the formulations.
2. Has history of seizure of any etiology, or of predisposition to seizures.
3. Has history of bulimia.
4. Has history of anorexia nervosa.
5. Has resting heart rate outside the normal range of 45 to 100 beats per minutes at Screening or Check-in (Day -1) and confirmed by a repeat measurement approximately 30 minutes following the initial measurement.
6. Has orthostatic blood pressure >=25 millimeter of mercury (mm Hg) at Screening or Check-in (Day -1) and confirmed by a repeat measurement approximately 30 minutes following the initial measurement.
7. Has sustained supine systolic blood pressure >=140 mm Hg or less than equal to (<=) 90 mm Hg or a diastolic blood pressure >=90 mm Hg or <=50 mm Hg at Screening or Check-in (Day -1) and confirmed by a repeat measurement approximately 30 minutes following the initial measurement.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration for Metformin Following a Single Dose of Metformin Administered Alone | Day 1: predose and at multiple timepoints (up to 48 hours) post-dose
Cmax: Maximum Observed Plasma Concentration of Metformin Following a Single Dose of Metformin and multiple Doses of naltrexone/bupropion | Day 14: predose and at multiple timepoints (up to 48 hours) post-dose
AUC(0-inf): Area Under the Plasma Concentration-time Curve from Time 0 to Infinity of Metformin Following a Single Dose of Metformin Administered Alone | Day 1: predose and at multiple timepoints (up to 48 hours) post-dose
AUC(0-inf): Area Under the Plasma Concentration-time Curve from Time 0 to Infinity of Metformin Following a Single Dose of Metformin and Multiple Doses of naltrexone/bupropion | Day 14: predose and at multiple timepoints (up to 48 hours) post-dose

SECONDARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration of bupropion, naltrexone and their metabolites (6beta-naltrexol, Bupropion, Hydroxybupropion, Threohydrobupropion, and Erythrohydrobupropion) following multiple doses of NB alone | Day 13 predose and at multiple timepoints (up to 12 hours) post-dose
Cmax: Maximum Observed Plasma Concentration of bupropion, naltrexone and their metabolites following multiple doses of naltrexone/bupropion and a single dose of metformin | Day 14: predose and at multiple timepoints (up to 12 hours) post-dose
AUC(0-tau): Area Under the Plasma Concentration-time Curve during a dosing interval for upropion, naltrexone and their metabolites (6beta-naltrexol, Bupropion, Hydroxybupropion, Threohydrobupropion, and Erythrohydrobupropion) | Day 13: predose and at multiple timepoints (up to 12 hours) post-dose for naltrexone/buprop alone, Day 14: predose and at multiple timepoints (up to 12 hours) post-dose, Day 14: predose and at multiple timepoints (up to 48 hours) post-dose
• Percentage of Participants who Experience at Least one Treatment Emergent Adverse Event (TEAE) | Day 1 upt to Day 45

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda